CLINICAL TRIAL: NCT04965181
Title: Mindfulness-based Smoking Cessation Enhanced With Mobile Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: University of Chicago (Other); University of Utah (Other); George Washington University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Claire Spears, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01CA237004 (NIH); R01CA237004 (NIH)
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully (Experimental): Participants will receive virtual group counseling based on the Mindfulness-Based Addiction Treatment (MBAT) group protocol, iQuit Mindfully text messages, and nicotine replacement therapy (NRT). MBAT consists of 8 weekly 2-hour sessions. NRT consists of 8 weeks of generic nicotine patches and nicotine lozenges. Participants who smoke >10 cigarettes/day will receive 4 weeks of 21 mg patches, 2 weeks of 14 mg patches, and 2 weeks of 7 mg patches. Those who smoke less than 10 cigarettes/day will receive 4 weeks of 14 mg patches and 4 weeks of 7 mg patches. Participants who smoke their first cigarette within 30 minutes of waking will receive 8 weeks of 4mg mini lozenges (6-9 4mg mini lozenges per day). Those who smoke their first cigarette over 30 minutes of waking will receive 8 weeks of 2mg mini lozenges (6-9 2mg mini lozenges per day). Participants will also be given the National Cancer Institute "Clearing the Air" booklet and a referral to the Tobacco Cessation Quitline.
  Interventions: Behavioral: Mindfulness-Based Addiction Treatment; Drug: Nicotine Replacement Therapy; Behavioral: Self-help materials; Behavioral: iQuit Mindfully
- iQuit Mindfully (Experimental): Participants will receive iQuit Mindfully text messages and nicotine replacement therapy (NRT). NRT consists of 8 weeks of generic nicotine patches and nicotine lozenges. Participants who smoke >10 cigarettes/day will receive 4 weeks of 21 mg patches, 2 weeks of 14 mg patches, and 2 weeks of 7 mg patches. Those who smoke less than 10 cigarettes/day will receive 4 weeks of 14 mg patches and 4 weeks of 7 mg patches. Participants who smoke their first cigarette within 30 minutes of waking will receive 8 weeks of 4mg mini lozenges (6-9 4mg mini lozenges per day). Those who smoke their first cigarette over 30 minutes of waking will receive 8 weeks of 2mg mini lozenges (6-9 2mg mini lozenges per day). Participants will also be given the National Cancer Institute "Clearing the Air" booklet and a referral to the Tobacco Cessation Quitline.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Self-help materials; Behavioral: iQuit Mindfully
- Mindfulness-based Addiction Treatment (MBAT) (Experimental): Participants will receive virtual group counseling based on the Mindfulness-Based Addiction Treatment (MBAT) group protocol and nicotine replacement therapy (NRT). MBAT consists of 8 weekly 2-hour sessions. NRT consists of 8 weeks of generic nicotine patches and nicotine lozenges. Participants who smoke >10 cigarettes/day will receive 4 weeks of 21 mg patches, 2 weeks of 14 mg patches, and 2 weeks of 7 mg patches. Those who smoke less than 10 cigarettes/day will receive 4 weeks of 14 mg patches and 4 weeks of 7 mg patches. Participants who smoke their first cigarette within 30 minutes of waking will receive 8 weeks of 4mg mini lozenges (6-9 4mg mini lozenges per day). Those who smoke their first cigarette over 30 minutes of waking will receive 8 weeks of 2mg mini lozenges (6-9 2mg mini lozenges per day). Participants will also be given the National Cancer Institute "Clearing the Air" booklet and a referral to the Tobacco Cessation Quitline.
  Interventions: Behavioral: Mindfulness-Based Addiction Treatment; Drug: Nicotine Replacement Therapy; Behavioral: Self-help materials
- Usual Care (Active Comparator): Participants in the usual care condition are provided with nicotine replacement therapy (NRT). NRT consists of 8 weeks of generic nicotine patches and nicotine lozenges. Participants who smoke >10 cigarettes/day will receive 4 weeks of 21 mg patches, 2 weeks of 14 mg patches, and 2 weeks of 7 mg patches. Those who smoke less than 10 cigarettes/day will receive 4 weeks of 14 mg patches and 4 weeks of 7 mg patches. Participants who smoke their first cigarette within 30 minutes of waking will receive 8 weeks of 4mg mini lozenges (6-9 4mg mini lozenges per day). Those who smoke their first cigarette over 30 minutes of waking will receive 8 weeks of 2mg mini lozenges (6-9 2mg mini lozenges per day). Participants will also be given the National Cancer Institute "Clearing the Air" booklet and a referral to the Tobacco Cessation Quitline.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Self-help materials

INTERVENTIONS:
Behavioral: Mindfulness-Based Addiction Treatment — Mindfulness-based Addiction Treatment (MBAT) consists of 8 weekly virtual 2-hour sessions that teach mindfulness and cognitive-behavioral strategies for smoking cessation.
  Other Names: MBAT
  Arms: Mindfulness-based Addiction Treatment (MBAT); Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully
Drug: Nicotine Replacement Therapy — Patch therapy (beginning quit day) for participants who smoke >10 cigarettes/day will consist of 4 weeks of 21 mg patches, 2 week of 14 mg patches, and 2 week of 7 mg patches. Patch therapy for participants who smoke less than 10 cigarettes/day will consist of 4 weeks of 14 mg patches and 4 weeks of 7 mg patches.
  Lozenge therapy (beginning quit day) for participants who smoke first cigarette within 30 minutes of waking up will consist of 8 weeks of 4mg lozenges. Lozenge therapy (beginning quit day) for participants who smoke first cigarette 30 minutes of more after they wake up will consist of 8 weeks of 2mg lozenges.
  Other Names: Generic Nicotine Patch; Generic Nicotine Lozenge
Behavioral: Self-help materials — Self-help materials for smoking cessation are based on the Treating Tobacco Use and Dependence Clinical Practice Guideline (Fiore et al., 2008) and include the "Clearing the Air" booklet developed by the National Cancer Institute (NCI) and a referral to the Tobacco Cessation Quitline (1-800-QUIT-NOW).
Behavioral: iQuit Mindfully — iQuit Mindfully involves text messages on each day between treatment sessions. The text messages provide mindfulness and cognitive-behavioral strategies and support for smoking cessation.
  Other Names: Mindfulness-based text messaging for smoking cessation
  Arms: Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully; iQuit Mindfully

SUMMARY:
The purpose of this study is to:

Aim I: Test the efficacy of a mindfulness-based text messaging program for smoking cessation ("iQuit Mindfully"), both as a standalone intervention and in combination with in-person counseling; and Aim II: Investigate the mechanisms through which mindfulness training impacts smoking cessation.

DETAILED DESCRIPTION:
This study is a 2 X 2 randomized controlled trial to investigate the effects of the iQuit Mindfully text messaging program, both as a standalone intervention and in combination with in-person counseling (Mindfulness-based Addiction Treatment; MBAT), compared to usual care. Participants will be randomized to one of four groups based on assignment to iQuit Mindfully text messages (yes/no) and in-person MBAT (yes/no):

* Usual Care (self-help materials + nicotine patch and nicotine lozenge treatment)
* MBAT (8 weekly virtual MBAT sessions + self-help materials + nicotine patch and nicotine lozenge treatment)
* iQuit Mindfully (iQuit Mindfully text messages + self-help materials + nicotine patch and nicotine lozenge treatment)
* MBAT + iQuit Mindfully (8 weekly virtual MBAT sessions + iQuit Mindfully text messages + self-help materials + nicotine patch and nicotine lozenge treatment)

All study participants will receive self-help smoking cessation materials, including the "Clearing the Air" booklet developed by the National Cancer Institute (NCI) and a referral to the Tobacco Cessation Quitline (1-800-QUIT-NOW). All study participants will also receive nicotine patches and lozenges. Assessments will occur at baseline and weeks 1, 3, 5, and 8. Follow-up assessments will occur at weeks 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current smoker with history of >3 cigarettes/day (and expired carbon monoxide [CO] >6ppm)
* motivated to quit within next 30 days
* valid home address in the greater Atlanta, GA area
* functioning telephone number
* can speak, read, and write in English

Exclusion Criteria:

* contraindication for nicotine patch or nicotine lozenge
* active substance abuse/dependence
* current suicidal ideation
* current use of tobacco cessation medications
* pregnancy, planning to become pregnant in the next 5 months, or lactation
* household member enrolled in the study
* enrolled in previous smoking cessation study based on mindfulness and/or text messaging at Georgia State University

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire A Spears, Ph.D, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Vidrine JI, Spears CA, Heppner WL, Reitzel LR, Marcus MT, Cinciripini PM, Waters AJ, Li Y, Nguyen NT, Cao Y, Tindle HA, Fine M, Safranek LV, Wetter DW. Efficacy of mindfulness-based addiction treatment (MBAT) for smoking cessation and lapse recovery: A randomized clinical trial. J Consult Clin Psychol. 2016 Sep;84(9):824-838. doi: 10.1037/ccp0000117. PMID 27213492
- [Derived] Spears CA, Mhende J, Hawkins C, Do VV, Hayat MJ, Eriksen MP, Hedeker D, Abroms LC, Wetter DW. Mindfulness-Based Smoking Cessation Delivered Through Telehealth and Text Messaging for Low-Income Smokers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Aug 1;11(8):e35688. doi: 10.2196/35688. PMID 35916707

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully | iQuit Mindfully | Mindfulness-based Addiction Treatment (MBAT) | Usual Care
Started | 141 | 146 | 147 | 70
Completed | 122 | 134 | 126 | 61
Not Completed | 19 | 12 | 21 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully | iQuit Mindfully | Mindfulness-based Addiction Treatment (MBAT) | Usual Care | Total
Number analyzed (Participants) | 141 | 146 | 147 | 70 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (12.8) | 49.8 (12.3) | 50.3 (13.1) | 53.0 (12.7) | 50.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 54 | 56 | 32 | 199
  Male | 84 | 92 | 91 | 38 | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 2 | 18
  Not Hispanic or Latino | 136 | 140 | 142 | 68 | 486
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 4 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 94 | 91 | 92 | 48 | 325
  White | 34 | 35 | 37 | 16 | 122
  More than one race | 6 | 13 | 6 | 1 | 26
  Unknown or Not Reported | 4 | 5 | 7 | 2 | 18
Cigarettes smoked per day at baseline [Mean (Standard Deviation); unit: Number of cigarettes per day] | 14.7 (7.3) | 15.4 (9.8) | 14.5 (7.5) | 13.6 (7.6) | 14.7 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Smoking Abstinence, 8 Weeks
Description: Self-report of not smoking any combustible tobacco products in the past 7 days (not even a puff), confirmed by expired carbon monoxide <6 ppm
Time Frame: 8 weeks after the start of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully: Participants receive virtual group counseling based on the Mindfulness-Based Addiction Treatment (MBAT) group protocol, iQuit Mindfully text messages, nicotine replacement therapy (NRT), and self-help materials in addition to regular check-in calls from the research team.
- iQuit Mindfully: Participants receive iQuit Mindfully text messages, nicotine replacement therapy (NRT), and self-help materials in addition to regular check-in calls from the research team.
- Mindfulness-based Addiction Treatment (MBAT): Participants receive virtual group counseling based on the Mindfulness-Based Addiction Treatment (MBAT) group protocol, nicotine replacement therapy (NRT), and self-help materials in addition to regular check-in calls from the research team.
- Usual Care: Participants in the usual care condition are provided with nicotine replacement therapy (NRT) and self-help materials, in addition to regular check-in calls from the research team.
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully | iQuit Mindfully | Mindfulness-based Addiction Treatment (MBAT) | Usual Care
Number analyzed (Participants) | 93 | 108 | 101 | 52
Participants | 13 | 29 | 26 | 12

2. Primary Outcome: Number of Participants With Confirmed Smoking Abstinence, 12 Weeks
Description: as for outcome 1
Time Frame: 12 weeks after the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully | iQuit Mindfully | Mindfulness-based Addiction Treatment (MBAT) | Usual Care
Number analyzed (Participants) | 107 | 123 | 110 | 55
Participants | 17 | 27 | 22 | 9

3. Primary Outcome: Number of Participants With Confirmed Smoking Abstinence, 24 Weeks
Description: Self-report of not smoking any combustible tobacco products in the past 7 days (not even a puff), confirmed by carbon monoxide < 6ppm and saliva cotinine < 20 ng/ml
Time Frame: 24 weeks after the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully | iQuit Mindfully | Mindfulness-based Addiction Treatment (MBAT) | Usual Care
Number analyzed (Participants) | 107 | 124 | 120 | 56
Participants | 18 | 22 | 16 | 8

4. Secondary Outcome: Home Mindfulness Practice (Number of Days Per Week)
Description: Self-reported frequency of home mindfulness practice (questionnaire; higher frequency means better outcome)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

5. Secondary Outcome: Dispositional Mindfulness (Mindful Attention Awareness Scale [MAAS])
Description: Self-reported dispositional mindfulness (questionnaire; higher frequency means better outcome; MAAS ranges 1-6)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

6. Secondary Outcome: Dispositional Mindfulness (Five Facet Mindfulness Questionnaire-Short Form [FFMQ-SF])
Description: Self-reported dispositional mindfulness (questionnaire; higher frequency means better outcome; FFMQ-SF ranges 24-120)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

7. Secondary Outcome: Self-compassion (Self-Compassion Scale-Short Form [SCS-SF])
Description: Self-reported self-compassion (questionnaire; higher frequency means better outcome; SCS-SF ranges 1-5)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

8. Secondary Outcome: Stress (Perceived Stress Scale [PSS])
Description: Self-reported stress (questionnaire; lower scores mean better outcome; PSS ranges 0-40)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

9. Secondary Outcome: Emotions (Positive and Negative Affect Schedule [PANAS])
Description: Self-reported positive and negative emotions (questionnaire; lower scores on PANAS-Negative Affect mean better outcome; higher scores on PANAS-Positive Affect mean better outcome; PANAS-Negative Affect and Positive Affect each range 10-50)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

10. Secondary Outcome: Craving and Withdrawal (Wisconsin Smoking Withdrawal Scale [WSWS])
Description: Self-reported craving and withdrawal (questionnaire; lower scores mean better outcome; subscale scores for each withdrawal symptom range 0-4)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

11. Secondary Outcome: Nicotine Dependence (Brief Wisconsin Dependence Motives Questionnaire [WISDM])
Description: Self-reported nicotine dependence (questionnaire; lower scores mean better outcome; subscale scores for each aspect of dependence range 1-7)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

12. Secondary Outcome: Self-efficacy (Self-Efficacy Scale)
Description: Self-reported self-efficacy to abstain from smoking (questionnaire; higher scores mean better outcome; subscale scores for managing positive affect, negative affect, and craving without smoking range 3-15)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

13. Secondary Outcome: Social Support (Multidimensional Scale of Perceived Social Support; Higher Scores Mean Better Outcome; Scores Range 1-7)
Description: Self-reported perceived social support (questionnaire)
Time Frame: During 8 weeks of treatment; 8, 12 and 24 weeks after the start of treatment
Reporting Status: Not Posted

14. Secondary Outcome: Program Evaluation (Questionnaire Developed for This Study to Evaluate Participants' Perceptions of the Helpfulness of Intervention Components, the Extent to Which They Would Recommend the Program to Others, and Suggestions for Improvement)
Description: Feedback about interventions and perceived benefits (questionnaire; for quantitative questions, higher scores mean better outcome; for questions about helpfulness and recommending to others, scores range 1-10; for perceived benefits of program, scores range 1-5)
Time Frame: 8 weeks after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events were assessed via regular check-in calls with participants.
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully | iQuit Mindfully | Mindfulness-based Addiction Treatment (MBAT) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/146 | 2/147 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/141 | 1/146 | 0/147 | 0/70
Other Adverse Events (participants affected / at risk) | 7/141 | 12/146 | 12/147 | 8/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully (N=141) | iQuit Mindfully (N=146) | Mindfulness-based Addiction Treatment (MBAT) (N=147) | Usual Care (N=70)
Severe disorientation (unrelated to study intervention) (Psychiatric disorders) | 0 | 1 | 0 | 0 — Participant was disoriented, likely due to substances consumed prior to study visit. Unrelated to study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness-based Addiction Treatment (MBAT) + iQuit Mindfully (N=141) | iQuit Mindfully (N=146) | Mindfulness-based Addiction Treatment (MBAT) (N=147) | Usual Care (N=70)
Mild side effects of nicotine replacement therapy (Product Issues) | 7 | 12 | 12 | 8 — Mild side effects of nicotine replacement therapy (e.g., itching, upset stomach)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT04965181/Prot_SAP_000.pdf